CLINICAL TRIAL: NCT05908045
Title: Have Physical Therapists Attitudes and Beliefs Towards Vital Assessment Changed Following the COVID-19 Pandemic?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Youngstown State University (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-294
Record Dates: First submitted 2023-06-15; First posted 2023-06-18 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Vital Signs
Keywords: vital sign; physical therapy; assessment; covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physical Therapists: Physical Therapists currently working in a clinical setting.
  Group Participants (Inclusion/Exclusion Criteria)
  Inclusion Criteria:
  1. Must be a licensed Physical Therapist
  2. Must be actively be involved in clinical practice
  3. Must have ≥ 5 years of experience practicing in a clinical setting as a Physical Therapist
  Exclusion Criteria:
  (1) Did not provide informed consent
  The survey will be disseminated across the American Physical Therapy Association (APTA) email lists. Further potential candidates may be identified through existing professional networks, clinical settings, and social medial/internet-based searching.
  Interventions: Other: KAP Survey

INTERVENTIONS:
Other: KAP Survey — This is a cross-sectional study that utilizes a KAP (knowledge, attitude, and practice) survey. This type of survey can be conducted on a representative sample of physical therapists who are currently involved in clinical practice. These types of surveys are useful for identifying gaps between what people know and how they act on that knowledge. There have been previous studies that have utilized KAP surveys when identifying knowledge, attitude, and practice behaviors of physical therapists.

SUMMARY:
Previous studies prior to the COVID-19 pandemic show that cardiovascular and blood pressure assessment by physical therapists is inadequate or lacking despite prior training. Since the COVID-19 pandemic, assessment of cardiovascular and respiratory function may become more critical as the manifestation of long COVID has become a concern. The purpose of this study is to determine whether physical therapists' attitudes and beliefs towards vital sign assessment have changed following the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a licensed Physical Therapist
2. Must be actively be involved in clinical practice
3. Must have ≥ 5 years of experience practicing in a clinical setting as a Physical Therapist

Exclusion Criteria:

(1) Did not provide informed consent

Ages: 23 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physical Therapists who are currently working in clinical practice that have a minimum of 5 years experience (based on ability to identify practice patterns prior to the COVID-19 pandemic).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
KAP Survey | Baseline
  The KAP Survey is divided into multiple sections (4 total) as outlined below:
  1. Demographic: Questions related to sample population (therapist) characteristics
  2. Prior COVID-19: Questions related to therapist attitudes and practices regarding vital assessment prior to COVID-19 pandemic.
  3. After COVID-19: Questions related to therapist attitudes and practices regarding vital assessment following COVID-19 pandemic.
  4. Knowledge: General knowledge questions related to vital assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Edmund C Ickert, PhD, Principal Investigator — Youngstown State University
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Severin R, Wang E, Wielechowski A, Phillips SA. Outpatient Physical Therapist Attitudes Toward and Behaviors in Cardiovascular Disease Screening: A National Survey. Phys Ther. 2019 Jul 1;99(7):833-848. doi: 10.1093/ptj/pzz042. PMID 30883642
- [Background] Albarrati AM PT, PhD. Outpatient physical therapy cardiovascular assessment: Physical therapist perspective and experience. Physiother Theory Pract. 2019 Sep;35(9):843-850. doi: 10.1080/09593985.2018.1458355. Epub 2018 Mar 29. PMID 29596007
- [Background] Faletra A, Bellin G, Dunning J, Fernandez-de-Las-Penas C, Pellicciari L, Brindisino F, Galeno E, Rossettini G, Maselli F, Severin R, Mourad F. Assessing cardiovascular parameters and risk factors in physical therapy practice: findings from a cross-sectional national survey and implication for clinical practice. BMC Musculoskelet Disord. 2022 Aug 4;23(1):749. doi: 10.1186/s12891-022-05696-w. PMID 35927658
- [Background] Frese EM, Richter RR, Burlis TV. Self-reported measurement of heart rate and blood pressure in patients by physical therapy clinical instructors. Phys Ther. 2002 Dec;82(12):1192-200. PMID 12444878